CLINICAL TRIAL: NCT01991743
Title: A Randomized Controlled Trial Comparing Combined Spinal- Epidural Dosing Strategies for External Cephalic Version
Brief Title: A Trial Comparing Combined Spinal- Epidural Dosing Strategies for External Cephalic Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Vice Chair Research Department of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00050371
Record Dates: First submitted 2013-10-29; First posted 2013-11-25 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy; Pain
Keywords: Version; Pregnancy; Vaginal Delivery; Pain Control; Combined Spinal Epidural
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Drug:Group 2.5 (Active Comparator): Administration of 2.5 mg bupivacaine
  Interventions: Drug: Group 2.5
- Group 5 (Active Comparator): Administration of 5 mg bupivacaine.
  Interventions: Drug: Group 5
- Group 7.5 (Active Comparator): Administration of 7.5mg bupivacaine.
  Interventions: Drug: Group 7.5
- Group 10 (Active Comparator): Administration of 10 mg bupivacaine.
  Interventions: Drug: Group 10

INTERVENTIONS:
Drug: Group 2.5 — Administration of bupivacaine 2.5 mg.
  Other Names: 2.5 mg bupivacaine
  Arms: Drug:Group 2.5
Drug: Group 5 — Administration of 5 mg bupivacaine
  Other Names: 5 mg bupivacaine
  Arms: Group 5
Drug: Group 7.5 — Administration of 7.5 mg bupivacaine
  Other Names: Administration of 7.5 mg bupivacaine.
  Arms: Group 7.5
Drug: Group 10 — Administration of 10mg bupivacaine.
  Other Names: Administration of 10mg bupivacaine.
  Arms: Group 10

SUMMARY:
We plan to conduct a prospective, single blinded, randomized clinical trial to assess the impact of combined spinal-epidural dosing on the success rate of, and patient satisfaction during, external version for breech fetal position and the incidence of vaginal vs. Cesarean delivery.

The research aim of this project is to determine the ideal neuraxial dosing strategy to maximize success of external cephalic version (ECV).

The research questions, does a combined spinal-epidural (CSE) of a higher dose result in greater success in converting a breech presentation to vertex during external cephalic version (ECV).

The hypotheses of this project is that CSE at higher dose will result in greater ECV success than analgesic dosing.

The research significance:Increasing the success and comfort of ECV for fetal malpresentation may help decrease the cesarean section rate.

DETAILED DESCRIPTION:
At term 2 to 3% of singleton pregnancies are in breech presentation. Many of these deliveries are managed by cesarean delivery due to higher neonatal morbidity associated with vaginal breech delivery. However, cesarean delivery, the safer option for the baby, is associated with a higher incidence of maternal complications for both the current and subsequent pregnancies. External cephalic version (ECV) is a procedure commonly used to attempt to manually rotate the fetus into vertex position. This facilitates vaginal delivery and thus avoids higher maternal and/or neonatal complications. (Hofmeyr Cochrane Review) Obstetricians generally perform versions after 36 weeks gestational age with a reportable success rate of 50-80%, depending on several factors, including patient characteristics. (Fortunato, Zhang, ACOG 1997 ECV) The most common technique involves external manipulation of the fetal position preceded by pharmacologic uterine relaxation. Until recently, pain relief was generally provided in the form of intravenous opioids such as fentanyl. A more efficacious form of analgesia is the use of neuraxial opioids and local anesthetics (neuraxial analgesia), a technique commonly used for labor and delivery analgesia.

Two non-randomized studies of neuraxial analgesia compared to systemic analgesia found improved success of external cephalic version in the neuraxial analgesia groups.(Carlan, Birnbach) Three randomized trials have conflicting results: 2 demonstrate an increase in success, one shows no difference. (Dugoff, Schorr, Mancuso) None of these studies have blinded the obstetrician performing the version. In 2010, Lavoie and colleagues completed a meta-analysis looking at ECV performed under analgesic and anesthetic neuraxial doses. The analgesic dose included spinal bupivacaine and epidural dosing. The anesthestic groups gave higher doses of spinal or epidural bupivacaine. This meta-analysis suggested that those patients who had received an anesthetic dose of had more successful ECV. All published studies examining pain outcomes have demonstrated that neuraxial analgesia results in greater patient comfort during this procedure.

The American College of Obstetricians and Gynecologists (ACOG) has stated, "Currently there is not enough evidence to make a recommendation favoring or opposing anesthesia during ECV (external cephalic version) attempts."

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients age 18 and older
* Breech presentation
* Singleton gestation .scheduled for ECV desiring CSE.

Exclusion Criteria:

* Refusal
* Contraindication to neuraxial (coagulopathy, anticoagulant use, local infection, sepsis etc) .Rupture of membranes.
* Drop-out: Patients may choose to drop-out of the study at any time. The physicians involved in this study may choose to end a patient's involvement in the study at their discretion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-05; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Study Director — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmeyr GJ. Interventions to help external cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2002;(2):CD000184. doi: 10.1002/14651858.CD000184. PMID 12076384
- [Background] Fortunato SJ, Mercer LJ, Guzick DS. External cephalic version with tocolysis: factors associated with success. Obstet Gynecol. 1988 Jul;72(1):59-62. PMID 3288930
- [Background] Zhang J, Bowes WA Jr, Fortney JA. Efficacy of external cephalic version: a review. Obstet Gynecol. 1993 Aug;82(2):306-12. PMID 8336883
- [Background] ACOG practice patterns. External cephalic version. Number 4, July 1997. American College of Obstetricians and Gynecologists. Int J Gynaecol Obstet. 1997 Oct;59(1):73-80. No abstract available. PMID 9359456
- [Background] Carlan SJ, Dent JM, Huckaby T, Whittington EC, Shaefer D. The effect of epidural anesthesia on safety and success of external cephalic version at term. Anesth Analg. 1994 Sep;79(3):525-8. doi: 10.1213/00000539-199409000-00021. PMID 8067558
- [Background] Birnbach DJ, Matut J, Stein DJ, Campagnuolo J, Drimbarean C, Grunebaum A, Kuroda MM, Thys DM. The effect of intrathecal analgesia on the success of external cephalic version. Anesth Analg. 2001 Aug;93(2):410-3, 4th contents page. doi: 10.1097/00000539-200108000-00035. PMID 11473871
- [Background] Dugoff L, Stamm CA, Jones OW 3rd, Mohling SI, Hawkins JL. The effect of spinal anesthesia on the success rate of external cephalic version: a randomized trial. Obstet Gynecol. 1999 Mar;93(3):345-9. doi: 10.1016/s0029-7844(98)00456-6. PMID 10074976
- [Background] Schorr SJ, Speights SE, Ross EL, Bofill JA, Rust OA, Norman PF, Morrison JC. A randomized trial of epidural anesthesia to improve external cephalic version success. Am J Obstet Gynecol. 1997 Nov;177(5):1133-7. doi: 10.1016/s0002-9378(97)70029-2. PMID 9396908
- [Background] Mancuso KM, Yancey MK, Murphy JA, Markenson GR. Epidural analgesia for cephalic version: a randomized trial. Obstet Gynecol. 2000 May;95(5):648-51. doi: 10.1016/s0029-7844(99)00611-0. PMID 10775722
- [Background] Lavoie A, Guay J. Anesthetic dose neuraxial blockade increases the success rate of external fetal version: a meta-analysis. Can J Anaesth. 2010 May;57(5):408-14. doi: 10.1007/s12630-010-9278-4. Epub 2010 Feb 3. PMID 20127530
- [Background] Sullivan JT, Grobman WA, Bauchat JR, Scavone BM, Grouper S, McCarthy RJ, Wong CA. A randomized controlled trial of the effect of combined spinal-epidural analgesia on the success of external cephalic version for breech presentation. Int J Obstet Anesth. 2009 Oct;18(4):328-34. doi: 10.1016/j.ijoa.2009.02.006. Epub 2009 Aug 13. PMID 19682886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 240 patients were enrolled and allocated to one of four bupivicaine dose groups
Period: Overall Study
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Started | 60 | 60 | 60 | 60
Completed | 60 | 60 | 59 | 60
Not Completed | 0 | 0 | 1 | 0
Not completed — external cephalic version not performed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10 | Total
Number analyzed (Participants) | 60 | 60 | 59 | 60 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 59 | 60 | 239
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 60 | 60 | 59 | 60 | 239
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 59 | 60 | 239
  Male | 0 | 0 | 0 | 0 | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m^2, resulting from mass in kilograms and height in meters.
  kg/m^2 | 29 [25 to 32] | 27 [26 to 30] | 28 [26 to 30] | 29 [26 to 32] | 28.5 [25 to 32]
Estimated Gestational Age [Median (Inter-Quartile Range); unit: days] | 263 [260 to 266] | 261 [259 to 265] | 261 [259 to 264] | 261 [259 to 266] | 261 [259 to 266]
Duration of Procedure [Median (Inter-Quartile Range); unit: minutes] | 7 [4 to 15] | 7 [4 to 14] | 11 [5 to 17] | 8 [4 to 15] | 7 [4 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of External Cephalic Version
Description: Rates of successful version evaluated among the 4 dose groups.
Time Frame: Completion of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Number analyzed (Participants) | 60 | 60 | 59 | 60
Participants | 31 | 31 | 31 | 30

2. Secondary Outcome: Mode of Delivery
Time Frame: To time of delivery
Measure: Number; unit: count of participants
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Number analyzed (Participants) | 60 | 60 | 59 | 60
count of participants
  Vaginal | 26 | 23 | 28 | 24
  Cesarean | 34 | 37 | 31 | 36

3. Secondary Outcome: Indication of Cesarean Delivery
Time Frame: To time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Number analyzed (Participants) | 60 | 60 | 59 | 60
Participants
  Malposition | 27 | 26 | 25 | 25
  Arrest of LAbor | 4 | 4 | 2 | 4
  Nonreassuring Fetal Status | 1 | 4 | 3 | 5
  Emergency | 2 | 3 | 1 | 2

4. Secondary Outcome: Pain Score During the Procedure
Description: pain score during the procedure (Visual Analog Score: VAS=0 no pain -100 worst pain imaginable, scale)
Time Frame: < 20 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Number analyzed (Participants) | 60 | 60 | 59 | 60
units on a scale | 12 [3 to 25] | 5 [1 to 18] | 4 [0 to 9] | 4 [0 to 10]

5. Secondary Outcome: Abdominal Relaxation
Description: Obstetrician rating of participants abdominal relaxation (Visual analog score: VAS score= 0 no relaxation- complete relaxation 100)
Time Frame: <20 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Drug:Group 2.5 | Group 5 | Group 7.5 | Group 10
Number analyzed (Participants) | 60 | 60 | 59 | 60
units on a scale | 78 [63 to 91] | 83 [71 to 92] | 84 [77 to 94] | 88 [73 to 95]

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- Group 2.5: Bupivicaine 2.5 mg
- Group 5: Bupivicaine 5 mg
- Group 7.5: Bupivicaine 7.5 mg
- Group 10: Bupivicaine 10 mg
Arm/Group | Group 2.5 | Group 5 | Group 7.5 | Group 10
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
The limitations include group allocation concealment and lack of a control group. The obstetrician's assessment of success, pain, anxiety, and fetus status may have prejudiced the decision to proceed or persist with external cephalic version.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No